CLINICAL TRIAL: NCT04765267
Title: Evaluation of Micronutrients With Topical Corticosteroid Versus Topical Corticosteroid in Management of Symptomatic Oral Lichen Planus: Three-arm Randomized Clinical Trial
Brief Title: Micronutrients in Management of Symptomatic Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Shousha, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMED 3-7-2
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Oral Lichen Planus
Keywords: micronutrients; topical corticosteroids
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Zinc Sulfate; Cholecalciferol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical Corticosteroid with Systemic Zinc. (Active Comparator): Octozinc: Zinc sulphate heptahydrate 25 mg tablets - October Pharma
  Interventions: Dietary Supplement: Zinc sulphate heptahydrate
- Topical Corticosteroid with Systemic Vitamin D (Active Comparator): Cholecalciferol: vitamin D3 15 ml oral solution - Medical Union Pharmaceuticals
  Interventions: Dietary Supplement: Zinc sulphate heptahydrate
- Topical Corticosteroid (Other): Kenacort A Orabase: triamcinolone acetonide 0.1% adhesive paste - Dermapharm
  Interventions: Dietary Supplement: Zinc sulphate heptahydrate

INTERVENTIONS:
Dietary Supplement: Zinc sulphate heptahydrate — Dietary supplements
  Other Names: Cholecalciferol: vitamin D3 oral solution

SUMMARY:
Treatment of oral lichen planus is challenging. Diverse therapeutic modalities have been suggested, but a permanent cure is not yet available. In some OLP patients, topical corticosteroid alone is not sufficiently enough, thus it may require a supplementation to augment its effect. Micronutrients are gaining more attention as therapeutic modalities in immunologic disorders. Researchers are recommended to conduct further clinical studies are to assess the role of these elements in management of OLP (Gholizadeh & Sheykhbahaei, 2020). Among the less visited micronutrients are zinc and vitamin D. This trial will assess their role in management of OLP.

DETAILED DESCRIPTION:
The enrolled patients will be divided randomly into three groups. One group will receive topical Corticosteroid (Kenacort A Orabase: triamcinolone acetonide 0.1% adhesive paste - Dermapharm) four times daily, the second group will receive topical Corticosteroid (Kenacort A Orabase: triamcinolone acetonide 0.1% adhesive paste - Dermapharm) four times daily with systemic zinc (Octozinc: Zinc sulphate heptahydrate 25 mg tablets - October Pharma) twice daily and the third group will receive topical Corticosteroid (Kenacort A Orabase: triamcinolone acetonide 0.1% adhesive paste - Dermapharm) four times daily with systemic vitamin D (Cholecalciferol: vitamin D3 15 ml oral solution - Medical Union Pharmaceuticals) once daily. The patients will be recalled weekly for eight weeks. For every four weeks of topical corticosteroid application, topical oral antifungal (Daktarin 2% oral gel - miconazole) will be prescribed, four times daily for one week, to all the patients in the trial, to avoid secondary infection with oral candidiasis. The patients will be asked to prohibit the use of any topical or systemic medication during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from erosive or atrophic OLP
* Patients free from any visible oral lesions other than OLP.
* Patients who agreed to take the supplied interventions.
* Patient who will agree to participate in the study.
* Patients who will accept to sign the informed consent.

Exclusion Criteria:

* Patients suffering from any systemic disease.
* Treatment with any systemic treatment such as systemic steroids, other immunosuppressive drugs or non-steroidal anti-inflammatory drugs at least eight weeks.
* Treatment with any oral topical medications for at least four weeks prior to the study.
* Pregnant and lactating mothers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity | baseline (week 0), daily in week 1, week 1,week 2, week 3, week 4, week 5, week 6 and week 7
  Visual analogue scale (0-10)

SECONDARY OUTCOMES:
change in clinical improvement | baseline (week 0), week 1,week 2, week 3, week 4, week 5, week 6 and week 7
  measured using Thongprasom et al. scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aboushousha A, Kamal Y, Ali S. Supplementary zinc and vitamin D in management of symptomatic oral lichen planus: a three-arm randomized clinical trial. BMC Oral Health. 2025 Jun 2;25(1):872. doi: 10.1186/s12903-025-06173-1. PMID 40457259